CLINICAL TRIAL: NCT06644027
Title: Effect of Different Types of Disposable Absorbent Sheets on the Local Skin Microclimate and Incidence of Incontinence-associated Dermatitis in Patients With Incontinence in the ICU: a Multicenter Randomized Controlled Trial
Brief Title: Prevention of Incontinence-associated Dermatitis and Maintenance of Local Skin Microclimate：A Multicenter Study
Acronym: I-and-M-m
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sir Run Run Shaw Hospital (Other)
Collaborators: Shaoxing People's Hospital (Other); Jiangshan People's Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20240455
Record Dates: First submitted 2024-10-06; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Incontinence-associated Dermatitis
Keywords: incontinence-associated dermatitis; microclimate; Jefcare Sterile Medical Sheets

STUDY DESIGN:
Intervention Model Description: Experimental: Jefcare Sterile Medical Sheets Other: Molicare Premium Bed Mat
Masking Description: Wound Ostomy and Continence Specialist Nurses and Dermatologists; laboratory technician
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Molicare Premium Bed Mat (Other): Screening period (day 0): normal routine medical sheet and skin care regimen. Intervention days 1, 2, 3, 4, 5: MoliCare Premium Bed Mats and skin care regimen.
  Interventions: Device: Molicare Premium Bed Mat
- Jefcare Sterile Medical Sheets (Experimental): Screening period (day 0): normal routine medical sheet and skin care regimen. Intervention days 1, 2, 3, 4, 5: Jefcare Sterile Medical Sheets and skin care regimen.
  Interventions: Device: Jefcare Sterile Medical Sheets

INTERVENTIONS:
Device: Jefcare Sterile Medical Sheets — Screening period (day 0): normal routine medical sheet and skin care regimen. Intervention days 1, 2, 3, 4, 5: Jefcare Sterile Medical Sheets and skin care regimen.
  Arms: Jefcare Sterile Medical Sheets
Device: Molicare Premium Bed Mat — Screening period (day 0): normal routine medical sheet and skin care regimen. Intervention days 1, 2, 3, 4, 5: MoliCare Premium Bed Mats and skin care regimen.
  Arms: Molicare Premium Bed Mat

SUMMARY:
To explore the feasibility of Jefcare Sterile Medical Sheets in preventing incontinence-associated dermatitis and maintaining a stable local skin microclimate in adult patients in the intensive care unit.

DETAILED DESCRIPTION:
Jefcare Sterile Medical Sheet is an incontinence care product designed by researchers following the Expert consensus on the clinical application of disposable absorbent care products for adults with incontinence. The product has good laboratory test indicators and has the potential to prevent incontinence-associated dermatitis and maintain the stability of the local skin microclimate. Still, there is a lack of high-quality clinical studies.

ELIGIBILITY:
Inclusion Criteria:

1. Intensive care unit incontinent patients (incontinence time ≥2 days)
2. Age ≥18 years
3. patients at high risk of IAD (Perineal Assessment Tool ≥ 7)
4. Voluntarily participate in the study and sign an informed consent form. If the subject is unable to read and sign the informed consent form due to incapacitation or other reasons, their guardian is required to represent the informed process and sign the informed consent form. If the subject is unable to read the informed consent form (e.g., illiterate subjects), a witness will be required to witness the informed process and sign the informed consent form.

Exclusion Criteria:

1. Patients who have developed IAD
2. Expected subsequent stay in the intensive care unit <5 days
3. Use of nappies, pull-ups, incontinence pads, etc.
4. Simple urinary incontinence with indwelling catheterization, external urinary bag without leakage; simple fecal incontinence with built-in drainage device, external ostomy bag, OB tampon without leakage; double incontinence with indwelling catheterization, external urinary bag, built-in drainage device, external ostomy bag, OB tampon without leakage.
5. The IAD may affect the skin area within the scope of the disease that affects the IAD judgment.
6. The IAD may affect the skin area within the scope of the skin breaks, infection
7. Patients who are not suitable for turning and cannot tolerate the side-lying position.
8. Patients with known allergies or keloid scarring
9. Women who are known to be pregnant or breastfeeding or who are planning to have a baby during the study period.
10. Patients who have participated in a clinical trial of another drug or medical device within 3 months.
11. Patients who, in the opinion of the investigator, are not suitable for participation in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2024-10-10 (Estimated); Primary Completion 2025-04-10 (Estimated); Study Completion 2025-04-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of IAD | Follow-up on Day 2, Day 3, Day 4, and Day 5 of the intervention until the start of the IAD/end of the study i.e. day 5 of the intervention.
  incidence of IAD = number of cases of patients with IAD in the group/total number of patients in the group × 100%.

SECONDARY OUTCOMES:
The time of IAD occurrence | Follow-up on Day 2, Day 3, Day 4, and Day 5 of the intervention until the start of the IAD/end of the study i.e. day 5 of the intervention.
  Time to IAD after enrolment
The site and severity of IAD occurrence | Follow-up on Day 2, Day 3, Day 4, and Day 5 of the intervention until the start of the IAD/end of the study i.e. day 5 of the intervention
  IAD may affect a range of 14 skin regions. A patient was considered to have IAD onset as long as the patient had IAD in 1 place.
  Using the IAD categorization tool, the tool classifies the severity of IAD into 3 levels. level 0 is represented by intact skin, no redness, and no difference in comparison to the skin of other body parts. level 1 is represented by red, intact, and possibly erythematous skin with edema. level 2 is represented by red, broken, and possibly skin with edema, blisters, blisters, vesicles, eruption of the skin, excoriation, and infected skin.
The skin microclimate and skin barrier function | Total 2 times. 1 prior to intervention, 1 on occurrence of IAD or end of the study i.e. day 5 of the intervention.
  Examination site: 3cm below the belly button；the lower abdomen/pubic arch; the inner right thigh; the inner left thigh ; the lower left buttock; the lower right buttock.
  Examination indicators: Skin temperature , skin hydration, skin PH , melanin , erythema , transepidermal water loss. Three measurements were taken at each site and averaged.
The skin microclimate and skin barrier function | Total 2 times. 1 prior to intervention, 1 on occurrence of IAD or end of the study i.e. day 5 of the intervention.
  Examination indicators: Temperature of sheets
Date of faecal incontinence (post-intervention);Mean number of faecal incontinence per day (post-intervention). | The average number of medical sheets used per day:Follow-up on Day 2, Day 3, Day 4, and Day 5 of the intervention until the start of the IAD/end of the study i.e. day 5 of the intervention.
  Date of fecal incontinence (post-intervention) = total number of days of fecal incontinence post-intervention.
  Date of faecal incontinence (post-intervention) = Total number of fecal incontinence episodes post-intervention/total number of days of fecal incontinence post-intervention.
Average daily cost-effectiveness of medical sheets. | The average number of medical sheets used per day:Follow-up on Day 2, Day 3, Day 4, and Day 5 of the intervention until the start of the IAD/end of the study i.e. day 5 of the intervention.
  Average daily cost-effectiveness of medical sheets = average daily number of medical sheets used x cost of individual medical sheet.
Mycological examination | Total 2 times. 1 prior to intervention, 1 on occurrence of IAD or end of study i.e. day 5 of the intervention.
  A cotton swab impregnated with saline sampling solution was applied to the local skin in a circular pattern from the upper left buttock, gluteal cleft, upper right buttock, lower right buttock, posterior right thigh, posterior left thigh, lower left buttock, and perineum in a sequential order, and the sampling cotton swabs were rotated accordingly, and the swabs were applied to the culture medium after sampling. Then to the front of the patient, a cotton swab was taken in a circular pattern from the lower abdomen/pubic arch, the left inguinal fold between the genitals and the thighs, the left inner thigh, the right inner thigh, the right inguinal fold between the genitals and the right thigh, and the genitals in the order of applying a localized skin and the subsequent rotation of the sampling cotton swab, and the swabs were applied to the culture medium after sampling. Observe for fungal growth and multiplication within the medium.

CONTACTS AND LOCATIONS:
Overall Officials: hongyang Hu, Study Chair — Sir Run Run Shaw Hospital

IPD SHARING:
Plan to Share IPD: No